CLINICAL TRIAL: NCT07056712
Title: Effect of Fenugreek Seed Administration on the Components of Metabolic Syndrome, Insulin Sensitivity, and Insulin Secretion
Brief Title: Effect of Fenugreek Seed Administration on Metabolic Syndrome, Insulin Sensitivity, and Insulin Secretion
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Guadalajara (Other)
Responsible Party: Principal Investigator, Marisol Cortez Navarrete, Principal investigator, University of Guadalajara
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Fenugreek-MS
Record Dates: First submitted 2025-06-29; First posted 2025-07-09 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-06

CONDITIONS: Metabolic Syndrome
Keywords: Metabolic Syndrome; Fenugreek; Insulin Secretion; Insulin Sensitivity; Nutraceutic
MeSH Terms: conditions — Metabolic Syndrome; Insulin Resistance | interventions — fenugreek seed meal

STUDY DESIGN:
Intervention Model Description: A randomized, double-blind, placebo-controlled clinical trial
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fenugreek seed (Experimental): 500 mg of fenugreek seed before each meal for 12 weeks
  Interventions: Dietary Supplement: Fenugreek seed
- Placebo (Placebo Comparator): 500 mg of calcined magnesia before each meal for 12 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Fenugreek seed — Fenugreek seed: 1500 mg per day for 12 weeks
  Other Names: Trigonella foenum-graecum
  Arms: Fenugreek seed
Other: Placebo — Placebo: Calcined magnesia 1500 mg per day for 12 weeks
  Other Names: Calcined magnesia
  Arms: Placebo

SUMMARY:
Fenugreek has been shown to have beneficial effects on various metabolic abnormalities associated with metabolic syndrome (MS). However, no clinical trials have evaluated its effect on all components of MS, insulin sensitivity, and insulin secretion. Therefore, the main objective of this study is to assess the effect of fenugreek seed administration versus placebo on the components of metabolic syndrome, insulin sensitivity, and insulin secretion.

DETAILED DESCRIPTION:
A randomized, double-blind, placebo controlled clinical trial will be conducted in 28 patients with metabolic syndrome according to the criteria of the International Diabetes Federation. Patients will be assigned to two different arms: one group will receive fenugreek seed extract (1500 mg/day) or a matched placebo for 12 weeks.

At the beginning and end of the intervention, the following measurements will be taken: body weight, body mass index, waist circumference, body fat percentage, systolic blood pressure, diastolic blood pressure, glucose, triglycerides, total cholesterol, high-density lipoprotein cholesterol, low-density lipoprotein cholesterol, very-low-density lipoprotein, insulin, creatinine, uric acid, alanine aminotransferase, and aspartate aminotransferase. In addition, insulin sensitivity and insulin secretion will be calculated. Written informed consent will be obtained from all volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between 30 and 60 years old.
* Diagnosis of Metabolic Syndrome (MS) according to the International Diabetes Federation (IDF) criteria.

Waist circumference ≥90 cm in men and ≥80 cm in women, plus the presence of two or more of the following criteria:

* Fasting glucose ≥100 mg/dL or previous diagnosis of type 2 diabetes.
* Systolic Blood Pressure ≥130 mmHg.
* Diastolic Blood Pressure ≥85 mmHg.
* Triglycerides ≥150 mg/dL.
* HDL cholesterol <40 mg/dL in men and <50 mg/dL in women.

  * Body Mass Index between 25.0 and 34.9 kg/m².
  * Stable weight during the 3 months prior to the start of the study (weight variation less than 10%).
  * Not receiving pharmacological treatment for any component of MS, insulin sensitivity, and/or insulin secretion.
  * Signed informed consent form.

Non-Inclusion Criteria:

* Suspected or confirmed pregnancy.
* Breastfeeding period.
* Fasting glucose ≥126 mg/dL.
* LDL cholesterol ≥155 mg/dL.
* Triglycerides ≥500 mg/dL.
* Systolic blood pressure ≥140 mmHg and diastolic blood pressure ≥90 mmHg.
* Use of medications and/or supplements known to influence the study variables.
* History of kidney, thyroid, liver disease, or ischemic heart disease.
* Active smoker.
* Not using an effective and stable contraceptive method.

Exclusion Criteria:

* Voluntary withdrawal of informed consent.
* Treatment adherence ≤80%.
* Occurrence of a serious adverse event.
* Loss to follow-up.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2026-09-15 (Estimated); Study Completion 2026-09-15 (Estimated)

PRIMARY OUTCOMES:
Waist Circumference (WC) | Baseline to week 12 (end of intervention)
  Waist Circumference (WC) is evaluated at baseline and after 12 weeks with a flexible tape in the midpoint between the lowest rib and the iliac crest
Systolic Blood Pressure (SBP) | Baseline to week 12 (end of intervention)
  Systolic Blood Pressure (SBP) is measured at baseline and after 12 weeks with a digital sphygmomanometer
Diastolic Blood Pressure (DBP) | Baseline to week 12 (end of intervention)
  Diastolic Blood Pressure (DBP) is measured at baseline and after 12 weeks with a digital sphygmomanometer
High Density Lipoprotein Cholesterol (HDL-c) | Baseline to week 12 (end of intervention)
  High Density Lipoprotein Cholestero (HDL-c) is evaluated at baseline and after 12 weeks with enzymatic/colorimetric techniques
Triglycerides (TG) | Baseline to week 12 (end of intervention)
  Triglycerides (TG) are evaluated at baseline and after 12 weeks with enzymatic/colorimetric techniques
Fasting Plasma Glucose (FPG) | Baseline to week 12 (end of intervention)
  Fasting Plasma Glucose (FPG) is evaluated at baseline and after 12 weeks with enzymatic/colorimetric techniques
Insulin Sensitivity (IS) | Baseline to week 12 (end of intervention)
  Insulin Sensitivity (IS) will be calculated at baseline and week 12 with Matsuda index to get insulin sensitivity
Total Insulin Secretion (TIS) | Baseline to week 12 (end of intervention)
  Total Insulin Secretion (TIS) will be calculated at baseline and week 12. It is the result of the ratio between the AUC of insulin in a 2-h OGTT and the AUC of glucose in a 2-h OGTT. It allows estimating the proportion of total insulin secretion in relation to plasma glucose concentration.
First Phase of Insulin Secretion (FPIS) | Baseline to week 12 (end of intervention)
  The First Phase if Insulin Secretion (FPIS) will be calculated at baseline and week 12 with Stumvoll index to get first phase of insulin secretion

SECONDARY OUTCOMES:
Body Weight (BW) | Baseline to week 12 (end of intervention)
  Body Weight (BW) is evaluated at baseline and after 12 weeks with an inbody 270
Body Mass Index (BMI) | Baseline to week 12 (end of intervention)
  Body Mass Index (BMI) is calculated at baseline and after 12 weeks with the Quetelet index formula
Body Fat Percentage (BF%) | Baseline to week 12 (end of intervention)
  Body Fat Percentage (BF%) will be measured at baseline and week 12 with a bioimpedance analysis
Total Cholesterol (TC) | Baseline to week 12 (end of intervention)
  Total Cholesterol (TC) is evaluated at baseline and after 12 weeks with enzymatic/colorimetric techniques
Low Density Lipoprotein Cholesterol (LDL-c) | Baseline to week 12 (end of intervention)
  Low Density Lipoprotein Cholesterol (LDL-c) level will be calculated at baseline and week 12 with Friedewald formula to get LDL-c level
Very Low Density Lipoprotein (VLDL) | Baseline to week 12 (end of intervention)
  Very Low Density Lipoprotein (VLDL) is calculated at baseline and after 12 weeks as triglycerides/5
Aspartate Aminotransferase (AST) | Baseline to week 12 (end of intervention)
  Aspartate Aminotransferase (AST) is evaluated at baseline and after 12 weeks with enzymatic/colorimetric techniques
Alanine Aminotransferase (ALT) | Baseline to week 12 (end of intervention)
  Alanine Aminotransferase (ALT) is evaluated at baseline and after 12 weeks with enzymatic/colorimetric techniques
Creatinine | Baseline to week 12 (end of intervention)
  Creatinine is evaluated at baseline and after 12 weeks with enzymatic/colorimetric techniques
Uric Acid (UA) | Baseline to week 12 (end of intervention)
  Uric Acid (UA) is evaluated at baseline and after 12 weeks with enzymatic-colorimetric techniques
Adverse Events (AE) | Baseline to week 12 (end of intervention)
  Adverse Events (AE) of fenugreek seed or placebo will be identified by clinical evaluation from baseline week to week 12 with continuous surveillance

CONTACTS AND LOCATIONS:
Overall Officials: Marisol Cortez Navarrete, PhD, Principal Investigator — Institute of Experimental and Clinical Therapeutics (INTEC), CUCS, University of Guadalajara
Locations (1):
- Instituto de Terapéutica Experimental y Clínica (INTEC), Centro Universitario de Ciencias de la Salud (CUCS), Universidad de Guadalajara., Guadalajara, Jalisco, Mexico